CLINICAL TRIAL: NCT07162948
Title: The ICU-Recover Box: Using Smart Technology for Monitoring Health Status After ICU Admission Pilot Study 2.0
Brief Title: ICU-Recover Box 2.0, Smart Technology for Home Monitoring of ICU Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Sesmu M. Arbous, MD PhD MSc, professor dr MS Arbous, anesthesiologist-intensivist, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL86464.058.24
Record Dates: First submitted 2025-06-25; First posted 2025-09-09 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: ICU Acquired Weakness
Keywords: smart technology; post-ICU recovery; post intensive care syndrome; health care utilization; health related quality of life
MeSH Terms: conditions — postintensive care syndrome; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: The primary objective of this pilot study is to assess the feasibility of the use of smart technology, i.e. Corsano CardioWatch 287-2 and blood pressure monitor assembled in the so-called ICU-Recover Box, by persons that have been discharged from the ICU in the one year following hospital discharge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients receiving the ICU-recover box containing home monitoring devices (Other): Treatment of subjects on the ICU and on the ward will be conform current practice, protocols and guidelines.
  Patients discharged from the ICU will receive an ICU-Recover Box on one of the clinical wards of the LUMC filled with the Corsano CardioWatch 287-2 and a Corsano blood pressure cuff after they have given informed consent. Descriptions of the Corsano CardioWatch 287-2 and the blood pressure cuff are given in further detail in section 6 of this protocol.
  Patients will also be asked to answer three short questionnaires regularly via telephone namely the ICU-CONTENT short (37 items), health care utilization questionnaire and the user friendliness questionnaire.
  Interventions: Device: The ICU-Recover Box: using smart technology for monitoring health status after ICU admission Pilot 2.0

INTERVENTIONS:
Device: The ICU-Recover Box: using smart technology for monitoring health status after ICU admission Pilot 2.0 — The Corsano CardioWatch 287-2 measures blood pressure, heart rate, heart rate variability, respiratory rate, peripheral oxygen saturation, body temperature and their daily activity.This devices is used for personal management, never to directly base a diagnosis or treatment on. The patient has to download the Corsano App on his/her mobile phone.

SUMMARY:
Smart technology could improve quality of care in patients who have been admitted to the ICU and have been discharged from ICU and hospital, by early diagnosis of complications and early (ambulatory) treatment.

With the ICU-Recover Box and its smart technology the investigators see new opportunities to improve patient health and to recognize early if escalation of medical care is needed.

The primary objective of the pilot study is to assess the feasibility of the use of smart technology by persons that have been discharged from the ICU in the twelve months following ICU discharge.

DETAILED DESCRIPTION:
Rationale: Smart technology could improve quality of care in patients who have been admitted to the ICU and have been discharged from ICU and hospital, by early diagnosis of complications and early (ambulatory) treatment.

In times of increasing medical care consumption leading to increasing health care costs one has to adopt new ways of acquiring patient-specific knowledge and new ways of delivering care. To obtain this level of insight one needs a smart and connected health care system. With the ICU-Recover Box and its smart technology the investigators see new opportunities to improve patient health and to recognize early if escalation of medical care is needed. By intervening early, one can possibly improve the quality of life for a patient and reduce costs by reducing health care utilization.

Objectives: The primary objective of the pilot study is to assess the feasibility of the use of smart technology by persons that have been discharged from the ICU in the twelve months following ICU discharge. If this pilot study proves to be successful, smart technology will be used in future studies.

Study design: This is a single centre cohort study. Study population: The study population consists of 50 patients who have been discharged from the ICU Department to a general ward of the Leiden University Medical Centre.

Intervention: Patients who consent to take part in the study, receive an ICU-Recover Box on the general ward closely before hospital discharge. The ICU-Recover Box will contain the Corsano CardioWatch 287-2. This is a Conformité Européenne (CE)-marked wristwatch-sized medical device, designed to monitor a comprehensive array of vital parameters, blood pressure, heart rate, heart rate variability, respiratory rate, peripheral oxygen saturation, body temperature and their daily activity.. Results of any of the measurements will never be used for therapy or diagnosis. To calibrate the blood pressure function of the Corsano CardioWatch 287-2, the ICU-Recover Box will contain a blood pressure monitor. Furthermore, patients who take part in this study will be contacted at regular moments by phone (at 1, 2,3, 6, 9, and 12 months) for follow-up on quality of life, health care use, and satisfaction with the home monitoring device.

Main study parameters/endpoints: The primary endpoint of the study will be the feasibility of providing and following ICU patients with smart technology for twelve months after discharge from ICU of the Leiden University Medical Centre.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The Corsano CardioWatch 287-2 is Conformité Européenne (CE)-marked for medical use, non-invasive, easy-to-use and electrically safe within its intended use. Using this device is with very limited risks.

This study has some potential benefits for patients: first, patients can measure their own blood pressure, heart rate, heart rate variability, respiratory rate, peripheral oxygen saturation, body temperature and their daily activity. This can reassure patients and give them more insight in their own health (the so-called 'patient empowerment'). Furthermore, this data gives the doctor more insight in the health of patients. This might lead to early detection of infection, respiratory or circulatory insufficiency, and cognitive or mental impairment, but diagnoses are not directly based on measurements of the personal management devices. Patients will have their own responsibility for taking action in case of self-experienced deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been admitted to the ICU of the LUMC for > 24 hours.
* Patient has received mechanical ventilation.
* Patient masters the English or Dutch language.
* Patient is able to use smart technology at home. (i.e. Wi-Fi available, sufficient comprehension of smart technology).
* Patient can be contacted and informed about the ICU-Recover box on one of the clinical wards of the LUMC.
* Patient is discharged from a ward within the LUMC to home or an extra-hospital facility.

Exclusion Criteria:

* Patient is < 18 years old.
* Patient is pregnant.
* Patient breastfeeds during the course of the study.
* Patient is discharged for palliative care.
* Patient is considered an incapacitated adult.
* Patient is unwilling to sign the informed consent form.
* Patient is discharged to another hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Use of smart technology | 12 months
  · The percentage of included post-ICU patients that was able to use and actually did use smart technology for twelve consecutive months.
Acquisition of data | 12 months
  · That it was possible (y/n) to acquire the data from the remote monitoring and that the investigators were able to store and use the data for analyses

SECONDARY OUTCOMES:
Lessons Learnt | 12 months
  That the investigators have an inventory of the lessons learned and feedback from participants, collected by a predefined questionnaire. On a monthly base the investigators will contact participants and ask them: (1) 36 questions on quality of life; (2) 2 questions on health care utilization; and (3) 9 questions on the use of the Corsano equipment. The questions are customised and not part of standardised questionnaires. Some questions are open-ended, while some are scale based (almost never-almost always).
  The investigators will report the results of these questionnaires qualitatively, as no final "score" can be attributed to the filled out questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands